CLINICAL TRIAL: NCT00890604
Title: Outcomes Associated With the Application of the Normothermia Protocol in Patients With Severe Neurological Insult and Fever
Brief Title: Outcomes Associated With Application of a Normothermia Protocol in Patients With Severe Neurological Insult and Fever
Acronym: SNIF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Gaymar Industries, Inc. (Industry)
Responsible Party: Principal Investigator, Hilaire Thompson, Professor: School of Nursing, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 34140
Record Dates: First submitted 2009-04-28; First posted 2009-04-30 (Estimated); Last update posted 2024-01-30 (Actual); Status verified 2019-06

CONDITIONS: Subarachnoid Hemorrhage; Severe Traumatic Brain Injury
MeSH Terms: conditions — Subarachnoid Hemorrhage; Brain Injuries, Traumatic | interventions — Ibuprofen; Acetaminophen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard interventions for temperature control used in protocolized, stepwise fashion (Other): Normothermia Protocol- use of standard interventions in protocolized fashion (physical cooling, antipyretics)
  Interventions: Other: Stepwise normothermia protocol; Drug: Ibuprofen; Drug: Acetominophen
- Standard fever management/prevention interventions used in ad hoc fashion (No Intervention): standard interventions for fever prevention used in ad hoc fashion based on nurse decision making

INTERVENTIONS:
Other: Stepwise normothermia protocol — Use of standard care interventions in a protocolized/step-wise fashion instead of ad hoc based on nurse decision making which may include antipyretics, physical cooling measures.
  Arms: Standard interventions for temperature control used in protocolized, stepwise fashion
Drug: Ibuprofen — It is not the intent of the study to evaluate this drug but may be provided in conjunction with the Stepwise normothermia protocol.
  Arms: Standard interventions for temperature control used in protocolized, stepwise fashion
Drug: Acetominophen — It is not the intent of the study to evaluate this drug but may be provided in conjunction with the Stepwise normothermia protocol.
  Arms: Standard interventions for temperature control used in protocolized, stepwise fashion

SUMMARY:
When fever is present in patients with stroke, traumatic brain injury (TBI), or brain hemorrhage, it has been associated with worse outcomes including larger areas of tissue death, increased length of stay, worse degree of coma, lower ability to function, and higher mortality. Both adult and pediatric TBI national guidelines state that maintenance of normal body temperature should be a standard of care. However, no further standards or options are presented to specifically guide practice. The current ischemic stroke guidelines state that fever should be treated with fever-reducing agents and offer "cooling devices" as an option but do not provide specifics to guide practice. Over 50% of patients in the Neurosurgical Intensive Care Unit (ICU) at Harborview Medical Center develop fever during the course of their stay. With elevated temperatures the body consumes more oxygen than if the temperature was normal, causing less oxygen to be available to the brain. This may lead to injury of the brain cells and a diminished capacity for healing. Thus, temperature management in neurologically vulnerable patients is both a prevalent and problematic challenge. Based on this information the goal of the present proposal is to evaluate if 1) A standardized, step-wise approach to temperature management using a Normothermia Protocol is successful in achieving and maintaining normal temperature in Neurosurgical ICU patients; and 2) If maintenance of normal temperature will be associated with fewer episodes of diminished responsiveness in their neurological exams as evidenced by a measure of depth of coma, as measured by the Glasgow Coma Score (GCS) compared to a control group treated according to usual care.

ELIGIBILITY:
Inclusion Criteria:

1. Temperature > 38.3 Celsius
2. Meet brain injury criteria:

   * Traumatic brain injury with Glasgow Coma Scale score of 8 or less
   * Subarachnoid hemorrhage without vasospasm- Hunt and Hess grade III and below
   * Subarachnoid hemorrhage with vasospasm
3. First febrile episode
4. English speaking

Exclusion Criteria:

1. Skin breakdown
2. Bleeding disorders
3. Increased risk for clotting
4. Ongoing seizure activity
5. Allergy to medications used in the study
6. Prisoners
7. Pregnancy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2009-07 (Actual); Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Glasgow Coma Score | 24 hour

SECONDARY OUTCOMES:
temperature | hourly
length of stay (intensive care, hospital) | discharge

CONTACTS AND LOCATIONS:
Overall Officials: Brenda Everett, Principal Investigator — Harborview Injury Prevention and Research Center; Robin Hilier, Principal Investigator — Harborview Injury Prevention and Research Center
Locations (1):
- Harborview Medical Center, Seattle, Washington, United States